CLINICAL TRIAL: NCT00512993
Title: A Randomized, Multicenter, Open Phase III Study Comparing the Postoperative Use of Zoledronic Acid Versus no Treatment in Patients With Histological Tumor Residuals After Preoperative Anthracycline and Taxane Containing Chemotherapy for Primary Breast Cancer
Brief Title: Postoperative Use of Zoledronic Acid in Breast Cancer Patients After Neoadjuvant Chemotherapy
Acronym: NATAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Austrian Breast & Colorectal Cancer Study Group (Network); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 36; NATAN; ABCSG 29
Record Dates: First submitted 2007-08-03; First posted 2007-08-08 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Postoperative treatment with zoledronic acid; Preoperative anthracycline/taxane containing chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): Patients receive zoledronic acid (4mg) for 5 years. Additionally patients receive standard endocrine, radiologic and trastuzumab treatment, respectively
  Interventions: Drug: Zoledronic acid
- Observation (No Intervention): Patients will be under observation and receive standard endocrine, radiologic and trastuzumab treatment, respectively

INTERVENTIONS:
Drug: Zoledronic acid — Infusion of zoledronic acid (4 mg) every 4 weeks for six doses, followed by every 3 months for 8 doses, followed by every 6 months for 5 doses
  Other Names: Zometa
  Arms: Treatment

SUMMARY:
The purpose of this study is to determine the event-free survival (EFS) after zoledronic acid for 5 years versus no postoperative treatment in patients with "chemo-insensitive" breast cancer (ypT1-4 and/or ypN1-3) after preoperative anthracycline/taxane containing chemotherapy

DETAILED DESCRIPTION:
The study is restricted to patients having had primary systemic chemotherapy for stage II and III breast cancer. Participation in a preoperative chemotherapy trial investigating anthracycline and taxane based regimen is allowed, but not mandatory for all patients. Patients must have significant remaining tumor tissue in the breast and/or axillary lymph node. This implies resistance to further chemotherapy and a clinically relevant risk for relapse. Bisphosphonates have a distinct mechanism of action and have demonstrated efficacy in the treatment of breast cancer with metastasis to the bone as well as adjuvant treatment after surgery of primary breast cancer. The 3rd generation bisphosphonate zoledronic acid has a favorable toxicity profile and can be conveniently given to patients over a long term period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained and documented according to the local regulatory requirements prior to beginning specific protocol procedures;
* Complete baseline documentation sent to GBG;
* Prior preoperative chemotherapy for at least 4 cycles, of which at least two must contain a taxane and an anthracycline;
* Completely resected unilateral or bilateral primary carcinoma of the breast with histologically detectable tumor residuals (ypT1-4) and/or histology confirmed involvement of axillary nodes (ypN1-3). Sentinel node biopsy is allowed, but complete axillary clearance is mandatory in node positive cases;
* A maximum interval of 3 years from date of axillary surgery to entering this trial;
* Age 18 years or older;
* Karnofsky index >= 70%;
* Life expectancy of at least 10 years, disregarding the diagnosis of cancer;
* No clinical evidence of local recurrence or distant metastases. Complete staging work-up: All patients must have breast ultrasound, chest X-ray, ultrasound or CT scan of the liver within 3 months prior to registration, as well as (bilateral) mammography or breast MRI and bone scan within 8 months prior to registration. In case of a positive bone scan, bone X-ray is mandatory. Other tests may be performed as clinically indicated;
* Adequate renal and hepatic function (serum creatinine, bilirubin, and transaminases within 1.5 × upper normal range);
* Patients must be available and compliant for treatment and follow-up. Patients registered on this trial must be treated and followed up at the participating center.

Exclusion Criteria:

* Known hypersensitivity reaction to the investigational compound;
* Prior postoperative chemotherapy;
* Prior treatment with bisphosphonates since breast cancer surgery;
* Pregnant or lactating patients. Patients of childbearing potential must have a negative pregnancy test (urine or serum) within 14 days prior to registration and must implement adequate non-hormonal contraceptive measures (barrier methods, intra uterine contraceptive devices, sterilization) during study treatment;
* History of diseases with influence on bone metabolism, such as Paget's disease of bone and primary hyperparathyroidism or osteoporosis requiring treatment at the time of study entry or considered likely to become necessary within the six months
* Other serious illness or medical condition that may interfere with the understanding and giving of informed consent and the conduct of the study
* Prior or concomitant secondary malignancy (except non-melanomatous skin cancer or carcinoma in situ of the uterine cervix)
* Concurrent treatment with other experimental drugs or any other anti-cancer therapy;
* Abnormal renal function as evidenced by a calculated creatinine clearance < 30 ml/minute;
* Serum calcium concentration < 8.0 mg/dl (2.00 mmol/L) or > 12.0 mg/dl (3.00 mmol/L)
* Concurrent treatment with sex hormones. Prior treatment must be stopped before study entry;
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw, of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g.. extraction, implants)
* Male patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Estimated)
Dates: Start 2004-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The event-free survival (EFS) after zoledronic acid for 5 years versus no postoperative treatment in patients with "chemo-insensitive" breast cancer (ypT1-4 and/or ypN1-3) after preoperative anthracycline/taxane containing chemotherapy. | 5 years

SECONDARY OUTCOMES:
The overall survival in both treatment arms. | 5 years
The EFS with respect to the interval between surgery and randomization. | 5 years
The bone-metastasis free-survival in both arms. | 5 years
The toxicity of and compliance to zoledronic acid. | 5 years
The predictive value of primary breast tumor response on the effect of postoperative treatment. | 5 years
The prognostic impact of chemotherapy induced amenorrhea in premenopausal patients. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gunter von Minckwitz, Prof. MD, Study Chair — GBG Forschungs GmbH, Hessen, Germany; Peter Dubsky, MD, Study Chair — Austrian Breast & Colorectal Cancer Study Group
Locations (93):
- Austria (10):
  - A. ö. Krankenhaus der Barmherzigen Brüder, Interne Abteilung, Saint Veit A. D. Glan, Carinthia
  - Landeskrankenhaus Wolfsberg, Chirurgische Abteilung, Wolfsberg, Carinthia
  - Medizinische Universität Wien, Wien, Lower Austria
  - LKH Salzburg, Uni.klinik f. Innere Med. III/Onkol. Amb., Salzburg, Salzburg
  - LKH-Univ. Klinikum Graz, Onkologie, Graz, Styria
  - Universitäts Klinikum Innsbruck, Innsbruck, Tyrol
  - Allgemeines Krankenhaus der Stadt Linz, Innere Medizin 3/Zentrum f. Häm. u. Med. Onkologie, Linz, Upper Austria
  - Landeskrankenhaus Steyr, 2. Med. Abt. Onkologie, Steyr, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Abt. f. Innere Medizin IV, Wels, Upper Austria
  - Landeskrankenhaus Feldkirch, Rankweil, Vorarlberg
- Germany (83):
  - Ostalb-Klinikum, ABC Brustzentrum, Frauenklinik, Aalen, Baden-Wurttemberg
  - Klinikum Sindelfingen-Böblingen / Kliniken Böblingen, Frauenklinik, Böblingen, Baden-Wurttemberg
  - St. Vincentius Kliniken Karlsruhe, Karlsruhe, Baden-Wurttemberg
  - Onkol. Schwerpunktpraxis Dr. Knoblich, Loerrach, Baden-Wurttemberg
  - Universitätsklinikum Mannheim, Frauenklinik, Mannheim, Baden-Wurttemberg
  - Krankenhaus Siloah, Gynäkologie und Geburtshilfe, Pforzheim, Baden-Wurttemberg
  - Klinikum am Steinenberg, Reutlingen, Baden-Wurttemberg
  - Frauenklinik Rheinfelden, Rheinfelden, Baden-Wurttemberg
  - Krankenhaus Bad Cannstatt, Frauenklinik, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Frauenklinik, Tübingen, Baden-Wurttemberg
  - Kreiskrankenhaus Ebersberg, Gynäkologisch-onkologische Abteilung, Ebersberg, Bavaria
  - Universitätsklinikum Erlangen, Frauenklinik mit Poliklinik, Erlangen, Bavaria
  - Caritas-Krankenhaus St. Josef, Klinik für Frauenheilkunde und Geburtshilfe, Regensburg, Bavaria
  - Klinikum Rosenheim, Abt. Gynäkologie u. Geburtshilfe, Rosenheim, Bavaria
  - Praxis Dr. Gottschalk, Fachärztin für Frauenheilkunde und Geburtshilfe, Bernau bei Berlin, Brandenburg
  - Schwerpunktpraxis der Gynäkologie und Onkologie, Fürstenwalde, Brandenburg
  - Ruppiner Kliniken, Frauenklinik, Neuruppin, Brandenburg
  - Onkologische Schwerpunktpraxis, Bremen, City state Bremen
  - Evangelisches Diakonie-Krankenhaus, Frauenklinik, Bremen, City state Bremen
  - Facharzt für Frauenheilkunde und Geburtshilfe, Hamburg, Hamburg
  - Onkologie Bethanien, Onkologie / Tagesklinik, Frankfurt am Main, Hesse
  - St. Markus Krankenhaus, Frauenklinik, Frankfurt am Main, Hesse
  - Städt. Kliniken Frankfurt-Höchst, Frauenklinik, Frankfurt/Höchst, Hesse
  - Klinikum Stadt Hanau, Hanau, Hesse
  - Klinikum Kassel GmbH, Gynäkologische Ambulanz, Kassel, Hesse
  - Asklepios Klinik, Frauenklinik, Langen, Hesse
  - Asklepios-Klinik Lich, Frauenklinik, Lich, Hesse
  - St. Vincenz Krankenhaus, Frauenklinik, Limburg an der Lahn, Hesse
  - Universitätsklinikum, Frauenklinik / Mutter-Kind-Zentrum, Marburg, Hesse
  - GBG Forschungs GmbH, Neu-Isenburg, Hesse
  - St. Josefs-Hospital, Gynäkologie und Geburtshilfe, Wiesbaden, Hesse
  - Asklepios Paulinen Klinik, Frauenklinik, Wiesbaden, Hesse
  - Dr.-Horst-Schmidt-Kliniken GmbH, Klinik f. Gyn. und gyn. Onkologie, Wiesbaden, Hesse
  - Allgm. Krankenhaus Celle, Frauenklinik, Celle, Lower Saxony
  - Krankenhaus Cuxhaven, Frauenklinik, Cuxhaven, Lower Saxony
  - Kreiskrankenhaus Gifhorn, Interdisziplinäres Brustzentrum, Gifhorn, Lower Saxony
  - Onkologische Schwerpunktpraxis Dr. Tessen, Goslar, Lower Saxony
  - Kreiskrankenhaus Hameln, Brustzentrum, Hamelin, Lower Saxony
  - Henriettenstiftung, Hanover, Lower Saxony
  - Vinzenzkrankenhaus, Gynäkologie, Hanover, Lower Saxony
  - Gemeinschaftspraxis Gynäkologie, Hildesheim, Lower Saxony
  - Facharzt für Frauenheilkunde und Geburtshilfe, Ilsede, Lower Saxony
  - Schwerpunktpraxis, Internistisch-gynäkolog.-onkolog., Lüneburg, Lower Saxony
  - Klinikum Schaumburg, Kreiskrankenhaus Stadthagen, Gynäkologie und Geburtshilfe, Stadhagen, Lower Saxony
  - Universität Greifswald, Klinik für Frauenheilkunde und Geburtshilfe, Greifswald, Mecklenburg-Vorpommern
  - Dietrich-Bonhoeffer Klinikum, Frauenklinik, Neubrandenburg, Mecklenburg-Vorpommern
  - Klinikum Südstadt, Universitätsfrauenklinik, Rostock, Mecklenburg-Vorpommern
  - Onkologische Schwerpunktpraxis, Dres. Schäfer / Just / Görner, Bielefeld, North Rhine-Westphalia
  - Praxis für Innere Medizin, Hämatologie, internistische Onkologie, Bochum, North Rhine-Westphalia
  - Onkologische Schwerpunktpraxis Dr. Glados, Hämatologie / Internistische Onkologie, Coesfeld, North Rhine-Westphalia
  - Klinikum der Universität zu Köln, Klinik und Poliklinik für Gyn. und Geburtshilfe, Cologne, North Rhine-Westphalia
  - Klinikum der Universität zu Köln, Cologne, North Rhine-Westphalia
  - St. Elisabeth-KKH, Brustzentrum Koeln-Hohenlind, Cologne, North Rhine-Westphalia
  - Luisenkrankenhaus, Senologie, Brustzentrum, Düsseldorf, North Rhine-Westphalia
  - Hermann-Josef Krankenhaus, Frauenklinik, Erkelenz, North Rhine-Westphalia
  - St. Antonius Hospital, Klinik für Hämatologie u. Onkologie, Eschweiler, North Rhine-Westphalia
  - Universitätsklinikum Essen, Klinik für Frauenheilkunde und Geburtshilfe, Essen, North Rhine-Westphalia
  - Gynäkologische Praxis Dr. Deertz, Essen, North Rhine-Westphalia
  - Alfried-Krupp-Krankenhaus, Frauenklinik, Essen, North Rhine-Westphalia
  - Marienhospital Altenessen, Essen, North Rhine-Westphalia
  - Marienhospital Herne, Onkologische / Hämatologische Ambulanz, Herne, North Rhine-Westphalia
  - Elisabeth-Hospital, Frauenklinik, Ibbenbueren, North Rhine-Westphalia
  - Marienhospital Witten, Brustzentrum, Witten, North Rhine-Westphalia
  - St. Vincenz und Elisabeth-Hospital, Mainz, Rhineland-Palatinate
  - Uniklinikum, Klinik für Geburtshilfe und Gynäkologie, Mainz, Rhineland-Palatinate
  - Krankenhaus Neunkirchen gGmbH, Frauenklinik, Neunkirchen, Saarland
  - Klinikum Chemnitz gGmbH, Frauenklinik, Chemnitz, Saxony
  - Gemeinschaftspraxis, Fachärzte für Innere Medizin, Hämatologie und Internistische Onkologie, Dresden, Saxony
  - Technische Universität Dresden, Dresden, Saxony
  - Krankenhaus St. Elisabeth und St. Barbara Halle, Klinik für Gynäkologie und Geburtshilfe, Halle, Saxony-Anhalt
  - Klinikum der Otto-v.-Guericke-Universität, Frauenklinik, Magdeburg, Saxony-Anhalt
  - Klinikum Quedlinburg, Frauenklinik, Quedlinburg, Saxony-Anhalt
  - Johanniter-Krankenhaus Genthin-Stendal GmbH, Frauenheilkunde und Geburtshilfe, Stendal, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Ostholstein Kliniken GmbH Klinik Oldenburg, Zentrum für Gynäkologie und Geburtshilfe Sana Kliniken Ostholstein, Oldenburg in Holstein, Schleswig-Holstein
  - Praxisklinik, Krebsheilkunde für Frauen / Brustzentrum, Berlin, State of Berlin
  - DRK Kliniken Köpenick, Frauenklinik, Berlin, State of Berlin
  - Schwerpunktpraxis Gynäkologie, Onkologie, Naturheilverfahren, Tempelhof, State of Berlin
  - SRH Wald-Klinikum Gera gGmbH, Brustzentrum Ostthüringen, Gera, Thuringia
  - Universitätsklinikum, Klinik für Frauenheilkunde und Geburtshilfe, Jena, Thuringia
  - Intern. Gemeinschaftspraxis, Friedrichshafen
  - Krankenhaus Salzwedel, Salzwedel

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- See also: Related Info — http://www.germanbreastgroup.de